CLINICAL TRIAL: NCT02853370
Title: Bendamustine and Rituximab for the Treatment of Splenic Marginal Zone Lymphoma. The International Extranodal Lymphoma Study Group (IELSG) 36 Phase II Prospective Study
Brief Title: Bendamustine and Rituximab for the Treatment of Splenic Marginal Zone Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IELSG 36
Record Dates: First submitted 2016-07-26; First posted 2016-08-02 (Estimated); Results first posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-05

CONDITIONS: Marginal Zone B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Bendamustine Hydrochloride; Rituximab

ARMS (1):
- Bendamustine and Rituximab (Experimental): Induction Phase (Cycle 1 to Cycle 3 ):
  Bendamustine 90 mg/sqm i.v. d1 & d2* Rituximab 375 mg/m2 i.v. d1**
  Extended Phase (Cycle 4 to Cycle 6):
  Bendamustine 90 mg/sqm i.v. d1 & d2* Rituximab 375 mg/m2 i.v. d1
  From Cycle 4 to Cycle 6, every 4 weeks, depending on the response after the first 3 Cycles
  *Or days 2-3 according to institutional/patient/physician preference
  **Administration of Rituximab during cycle 1 and cycle 2 can be postponed to day 8 or 14 in case of risk of tumor lysis syndrome (TLS)
  Interventions: Drug: Bendamustine and Rituximab

INTERVENTIONS:
Drug: Bendamustine and Rituximab

SUMMARY:
Splenic Marginal Zone Lymphoma (SMZL) is a well-defined low-grade B-cell lymphoma,considered as a rare neoplasm accounting for about 2% of all non-Hodgkin's lymphomas (NHL) and represents for most cases of otherwise unclassifiable chronic lymphoid B-cell cluster of differentiation antigen 5 (CD5)-lymphoproliferative disorders. SMZL is characterized by an almost exclusive involvement of the spleen and bone marrow and in about 25% of cases the disease pursues an aggressive course and most patients die of lymphoma progression within 3-4 years.

Retrospective studies have indicated that purine analogous achieved very high response rates in both naïve and pre-treated patients. Moreover, the introduction of the anti-cluster of differentiation antigen 20 (CD20) humanized antibody rituximab, either used alone or in combination with chemotherapy has been reported to be very effective in producing a rapid clearance of neoplastic cells.

DETAILED DESCRIPTION:
Prospective, multicenter, open-label, phase II study, designed to determine efficacy and safety of a Chemo-immunotherapy with the combination of bendamustine + rituximab in patients with splenic marginal zone lymphoma.

Study Population: previously untreated (except for splenectomy and/or antiviral therapy for Hepatitis C Virus (HCV) infection) and symptomatic Splenic Marginal Zone patients.

Objectives: evaluation of the efficacy and the safety of R-Bendamustine in symptomatic Splenic Marginal Zone Lymphoma patients.

Primary Objective: efficacy of R-Bendamustine measured by Complete Response rate. Complete response rate defined as regression to normal size on CT of organomegaly (spleen, liver, lymph nodes); normalization of the blood counts and no evidence of circulating clonal cells, and no evidence or minor (≤ 5%) Bone Marrow (BM) infiltration detected by immunohistochemistry (IHC).

Treatment: The R-Bendamustine regimen consisted of 28-day cycle. Patients achieving a complete response (CR) after 3 cycles received only one more cycle of R-Bendamustine, while those achieving a partial response (PR) received 3 additional cycles of R-Bendamustine; if less than PR patients were withdrawn from the study

ELIGIBILITY:
Inclusion Criteria:

* Initial diagnosis of CD20+ Splenic Marginal Zone Lymphoma morphology confirmed by histology, cytology, immunophenotype (chromosomal abnormalities by quantitative multiplex Polymerase Chain Reaction (PCR) of short fluorescent fragments (QMPSF) is optional) according to World Health Organization (WHO) 2008 classification of Lymphoma criteria or according to the recommendation of the Splenic Lymphoma Group for non splenectomized patient.

  1. If patients not splenectomised: diagnosis on bone marrow biopsy (histology and immunohistochemistry), and blood (cytology, immunophenotype), chromosomal abnormalities by QMPSF optional.
  2. If patients splenectomised diagnosis on spleen, bone marrow biopsy (histology and immunohistochemistry), and blood (cytology, immunophenotype) chromosomal abnormalities by QMPSF optional.
* No previous treatment with immunotherapy or chemotherapy or radiotherapy unless pretreatment by mono corticotherapy.
* Patients requiring a treatment with at least one of the following situation:

  1. Symptomatic SMZL in not splenectomized patients

     1. Bulky (arbitrarily defined as ≥6 cm below left costal margin) or progressive or painful splenomegaly, without enlarged lymphoadenopathy, with or without cytopenia, not eligible for splenectomy or not willing splenectomy
     2. One of the following symptomatic/progressive cytopenias: Hb <10 g/dL, or Plat <80.000/mm3, or ANC <1.000/mm3, whatever the reason (autoimmune or hypersplenism or bone marrow infiltration) not eligible for splenectomy or not willing splenectomy
     3. SMZL with enlarged lymphoadenopathy or involvement of extranodal sites with or without cytopenia
  2. Symptomatic disease in SMZL splenectomised patients with rapidly raising lymphocyte counts, development of lymphadenopathy or involvement of extranodal sites.
  3. SMZL with concomitant hepatitis C infection who have not responded or are relapsed after Interferon and/or Ribavirin.
* Clinically and/or radiologically confirmed measurable disease before treatment start.
* Aged ≥ 18 yo at time of initial diagnosis and ≤ 80 yo.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Minimum life expectancy of >6 months.
* Voluntary signed informed consent before performance of any study related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
* The following laboratory values at screening:

  1. Absolute neutrophil count (ANC) ≥1.000/mm3 and Platelets ≥100.000/mm3, unless these abnormalities are related to bone marrow infiltration or to hypersplenism.
  2. Aspartate transaminase (AST) ≤2 x upper limit of normal (ULN); Alanine transaminase (ALT) ≤2 x ULN; total bilirubin ≤1.5 x ULN.
  3. Creatinine clearance ≥ 10 ml/min (as calculated by the Cockcroft-Gault formula)

All patients must:

1. Agree to abstain from donating blood while taking study drug therapy and following discontinuation of study drug therapy.
2. Agree not to share study medication with another person.
3. Agree to use an adequate method of contraception for women of childbearing potential during the study treatment and until 12 months after the end of the study treatment.
4. Agree to use an adequate method of contraception for men during the study treatment and until 6 months after the end of the study treatment

Exclusion Criteria:

1. Any type of lymphoma other than SMZL.
2. Patients with proven biopsy of histological transformation.
3. Contraindication to any drug contained in the chemotherapy regimen.
4. Myocardial infarction during last 3 months or unstable coronary disease or uncontrolled chronic symptomatic congestive heart insufficiency NYHA III - IV.
5. Uncontrolled hypertension.
6. Uncontrolled diabetes mellitus as defined by the investigator.
7. Active systemic infection requiring treatment.
8. Previously known HIV positive serology.
9. Active hepatitis B virus infection (presence of antigen HBS+; in case of presence of antibody anti HBC+ and anti HBS+, controls should be organized according to guidelines of AASLD and l'EASL).
10. Active and previously untreated HCV infection.
11. Prior history of malignancies other than lymphoma within 3 years (except for complete resection of basal cell carcinoma, squamous cell carcinoma of the skin, or in situ malignancy). Patients previously diagnosed with prostate cancer are eligible if (1) their disease was T1-T2a, N0, M0, with a Gleason score </=7, and a prostate specific antigen(PSA) </=10 ng/mL prior to initial therapy, (2) they had definitive curative therapy (ie, prostatectomy or radiotherapy) >/=2 years before Day 1 of Cycle 1, and (3) at a minimum 2 years following therapy they had no clinical evidence of prostate cancer, and their PSA was undetectable if they underwent prostatectomy or <1 ng/mL if they did not undergo prostatectomy.
12. Major surgery within 30 days before the inclusion in the study
13. A positive Coombs test without haemolysis or an autoimmune hemolytic anemia is not an exclusion criterion.
14. Impaired renal function with creatinine clearance <10 ml/min.
15. Severe chronic obstructive pulmonary disease with hypoxemia.
16. Medical condition requiring long-term use (>1 months) of systemic corticosteroids.
17. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
18. Prior participation in another study with experimental drug during the last 4 months.
19. Pregnant or currently breast-feeding woman.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Iannitto, MD, Study Chair — Presidio ospedaliero G. Moscati; UOC di Ematologia - Taranto
Locations (30):
- France (12):
  - Créteil (Hôpital Henri Mondor), Créteil
  - Dijon (CHU de Dijon - Hôpital d'Enfants), Dijon
  - Grenoble cedex 9 (CHU Michallon), Grenoble
  - Le Kremlin Bicêtre (Hôpital Bicêtre), Le Kremlin-Bicêtre
  - Le Mans (C.H. Le Mans), Le Mans
  - Lille cedex (CHRU Lille - Hôpital Claude Huriez), Lille
  - Pierre Bénite, Lyon Sud
  - Vandoeuvre-les-Nancy cedex (CHU Brabois), Nancy
  - Nantes cedex 01 (CHU de Nantes - Hôtel Dieu), Nantes
  - Paris cedex 10 (Hôpital Saint-Louis), Paris
  - Pessac cedex (Centre François Magendie), Pessac
  - Rouen (Centre Henri Becquerel), Rouen
- Italy (18):
  - Ospedale Civile Ss. Antonio E Biagio, Alessandria
  - A.O. Universitaria Ospedali Riuniti - Ospedale Umberto I Di Ancona, Ancona
  - Ospedale Armando Businco, Cagliari
  - A.O. Universitaria S. Martino Di Genova, Genova
  - Irst - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori - Sede Di Meldola (Fc), Meldola
  - Irccs Fondazione Centro S. Raffaele Del Monte Tabor, Milan
  - A.O. Universitaria Policlinico Di Modena, Modena
  - A.O. "V. Cervello", Palermo
  - A.O. Universitaria Policlinico Giaccone, Palermo
  - A.O. Universitaria Di Parma, Parma
  - Ausl Di Piacenza, Piacenza
  - Ospedale S. Maria Delle Croci Di Di Ravenna, Ravenna
  - Ospedale Bianchi - Melacrino - Morelli, Reggio Calabria
  - Ospedale Di S. Maria Nuova-Irccs, Reggio Emilia
  - Irccs Centro Di Riferimento Oncologico Di Basilicata (Crob), Rionero Sannitico
  - Irccs Istituto Dermatologico S. Gallicano (Ifo), Roma
  - Azienda Ospedaliera "S. Maria", Terni
  - Ospedale Di Circolo E Fondazione Macchi, Varese

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment lasted from 03 December 2012 to 13 November 2014
Pre-assignment Details: 78 patients were screened and 56 patients were eligible: 16 patients were ineligible for unconfirmed diagnosis of SMZL, 3 for age >80 years, 1 for withdrawal of the Informed Consent, 1 for treatment not started and 1 urgent treatment needed.
Groups:
- Bendamustine and Rituximab: Induction Phase (Cycle 1 to Cycle 3 ):
  Bendamustine 90 mg/sqm i.v. d1 & d2 or d2 & d3 Rituximab 375 mg/m2 i.v. d1
  Extended Phase (Cycle 4 to Cycle 6):
  Bendamustine 90 mg/sqm i.v. d1 & d2 Rituximab 375 mg/m2 i.v. d1
Period: Overall Study
Arm/Group | Bendamustine and Rituximab
Started | 56
Completed | 45
Not Completed | 11
Not completed — Physician Decision | 1
Not completed — Lack of Efficacy | 2
Not completed — Death | 1
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Bendamustine and Rituximab
Number analyzed (Participants) | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 38
  France | 18
ECOG Performance Status [Count of Participants; unit: Participants] — WHO performance status scale:
  0 - Able to carry out all normal activity without restriction
  1. - Restricted in physically strenuous activity but ambulatory and able to carry out light work
  2. - Ambulatory and capable of all self-care but unable to carry out any work; up and about more than 50% of waking hours
  3. - Capable of only limited self-care; confined to bed or chair more than 50% of waking hours
  4. - Completely disabled; cannot carry on any self-care; totally confined to bed or chair
  Participants
    Grade 2 | 2
    Grade 0 - 1 | 51
    Not recorded | 3
Bone Marrow (BM) Involvement [Count of Participants; unit: Participants]
  BM Involvement | 56
  No BM Involvement | 0
Thoracic and / or abdominal lymphadenopathy [Count of Participants; unit: Participants]
  Thoracic and / or abdominal lymphadenopathy | 34
  No Thoracic and / or abdominal lymphadenopathy | 22
Extranodal Involvement [Count of Participants; unit: Participants]
  Extranodal Involvement | 2
  No Extranodal Involvement | 54
IIL Prognostic Score [Count of Participants; unit: Participants] — The Lymphoma Italian Intergroup (IIL) have proposed a clinical score based on three parameters:
  1. Haemoglobin < 12 gr/dL
  2. LDH > ULN
  3. Albumin < 3.5 gr/dL
  Score:
  Low Risk non adverse factor; Intermediate Risk 1 adverse factor; High Risk 2-3 adverse factors.
  Participants
    Low (0) | 22
    Intermediate (1) | 14
    High (2 - 3) | 19
    Not recorded | 1

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate (CRR)
Description: Percentage of patients with complete response. Complete response to be assessed by means of CT-scan, Immunophenotype in blood and bone marrow (PET-scan optional) Complete response (CR) requires the disappearance of all evidence of disease
  1. Regression to normal size on CT of organomegaly (splenomegaly, hepatomegaly and lymphoadenopathies)
  2. Normalization of the blood counts (Hb >12 g/dl; platelets >100.000/mm3; neutrophils >1.500/mm3 and no evidence of circulating clonal B-cells)
  3. No evidence or minor (<5%) BM infiltration detected by immunohistochemistry
Time Frame: At the end of treatment (After 24 weeks of treatment)
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Bendamustine and Rituximab
Number analyzed (Participants) | 56
Percentage of patients | 73 [60 to 84]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Percentage of patients with complete and partial response. Partial response (PR) requires regression of 50% or greater in the measurable disease manifestations and no new sites of disease.
  This should include: resolution or decrease in spleen size, improvement on cytopenias and resolution or decrease in lymphadenopathy if present. Bone Marrow should show a decrease in the level of lymphoid infiltration and improvement of the haemopoietic reserve
Time Frame: At the end of treatment (After 24 weeks of treatment)
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Groups:
- Bendamustine and Rituximab: Induction Phase (Cycle 1 to Cycle 3 ):
  Bendamustine 90 mg/sqm i.v. d1 & d2 or d2 & d3 Rituximab 375 mg/m2 i.v. d1**
  Extended Phase (Cycle 4 to Cycle 6):
  Bendamustine 90 mg/sqm i.v. d1 & d2 Rituximab 375 mg/m2 i.v. d1
Arm/Group | Bendamustine and Rituximab
Number analyzed (Participants) | 56
Percentage of patients | 91 [80 to 97]

3. Secondary Outcome: 3-year Progression Free Survival (PFS)
Description: Percentage of patients free from disease progression after 3 years from study entry.
  Progression is defined as reappearance of cytopenia or lymphoma relapse/ progression with enlarged lymph node(s) or spleen if present, histologic transformation or death as a result of any cause.
Time Frame: 3 years after study entry
Measure: Number (99% Confidence Interval); unit: Percentage of patients
Arm/Group | Bendamustine and Rituximab
Number analyzed (Participants) | 56
Percentage of patients | 90 [77 to 96]

4. Secondary Outcome: 3-years Duration of Response (DOR)
Description: Percentage of responding patients after 3 years from study entry. DOR is defined for all patients who achieved a response (CR and PR)
Time Frame: 3 years from study entry
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Bendamustine and Rituximab
Number analyzed (Participants) | 56
Percentage of patients | 93 [81 to 98]

5. Secondary Outcome: 3-years Event Free Survival (EFS)
Description: Percentage of patients free from events after 3 years from study entry. Events are defined as any treatment failure including disease progression, or discontinuation of treatment for any cause (eg, disease progression, toxicity, patient preference, initiation of new treatment without documented progression, or death).
Time Frame: 3 years after study entry
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Bendamustine and Rituximab
Number analyzed (Participants) | 56
Percentage of patients | 80 [65 to 89]

6. Secondary Outcome: 3-years Overall Survival Rate
Description: Percentage of patients alive after 3 years from study entry
Time Frame: 3 years after treatment start
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Bendamustine and Rituximab
Number analyzed (Participants) | 56
Percentage of patients | 96 [84 to 98]

7. Secondary Outcome: 5 Years Progression Free Survival (PFS) -
Description: Percentage of patients free from disease progression after 5 years from treatment start. Progression is defined as reappearance of cytopenia or lymphoma relapse/ progression with enlarged lymph node(s) or spleen if present, histologic transformation or death as a result of any cause.
Time Frame: Five years after study entry
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Bendamustine and Rituximab
Number analyzed (Participants) | 56
Percentage of patients | 83 [71 to 91]

8. Secondary Outcome: 5 Years Overall Survival (OS)
Description: Percentage of patients alive after 5 years from study entry
Time Frame: Five years after study entry
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Bendamustine and Rituximab
Number analyzed (Participants) | 56
Percentage of patients | 93 [82 to 97]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs): from the date of informed consent signature until 30 days after last treatment administration (8 months). Serious AEs suspected to be related to the study: until the end of study (5 years) .
Arm/Group | Bendamustine and Rituximab
All-Cause Mortality (participants affected / at risk) | 4/56
Serious Adverse Events (participants affected / at risk) | 14/56
Other Adverse Events (participants affected / at risk) | 50/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine and Rituximab (N=56)
Angioplasty (Surgical and medical procedures) | 1 (1)
Pancytopenia (Investigations) | 1 (1)
Malignant peripheral nerve sheath tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Coagulation disorders (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (2)
Paraneoplastic fever (General disorders) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine and Rituximab (N=56)
Anaemia (Blood and lymphatic system disorders) | 24 (42)
Leukopenia (Blood and lymphatic system disorders) | 28 (82)
Neutropenia (Blood and lymphatic system disorders) | 31 (98)
Thrombocytopenia (Blood and lymphatic system disorders) | 26 (51)
Investigations (Investigations) | 3 (4)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 4 (10)
Nervous system disorders (Nervous system disorders) | 3 (3)
General disorders and administration site conditions (General disorders) | 13 (22)
Gastrointestinal disorders (Gastrointestinal disorders) | 23 (37)
Skin disorder (Skin and subcutaneous tissue disorders) | 10 (19)
Infections (Infections and infestations) | 7 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/70/NCT02853370/Prot_SAP_000.pdf